CLINICAL TRIAL: NCT04700865
Title: The South-Norway Atrial Fibrillation Screening Study
Acronym: AFstudien
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sorlandet Hospital HF (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20/09000-7
Record Dates: First submitted 2020-12-26; First posted 2021-01-08 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2020-12

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Examination (Other): Continuous ECG monitoring for minimum 3 days
  Interventions: Diagnostic Test: AF screening

INTERVENTIONS:
Diagnostic Test: AF screening — Continous ECG monitoring for minimum 3 days

SUMMARY:
Atrial fibrillation (AF) is the most common sustained cardiac rhythm disorder. The most serious common complication of AF is ischemic stroke.The aim of this study is to investigate the yield of AF screening with a continuous ECG monitor (ECG247) and to estimate the prevalence of silent AF

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common sustained cardiac rhythm disorder. The most serious common complication of AF is ischemic stroke. Many AF cases are undiagnosed due to the asymptomatic and intermittent nature of AF (silent AF). Today there is no simple and inexpensive method of detecting silent AF and thus preventing stroke. The ECG247 Sensor is a new Norwegian digital clinical tool for out-of-hospital self-testing of AF. The innovation project has originated from the University of Agder and Sorlandet Hospital. The COVID19 pandemic is realizing more than ever the need for single-use self-testing out-of-hospital diagnostic tools.

The general aim of this open non-randomized study is to investigate the yield of AF screening with a continuous ECG monitor (ECG247) and to estimate the prevalence of silent AF in a cohort of 1500 65-year-old individuals with additional risk factors for stroke.

If the study results indicate that easy-to-use continuous AF-screening-devices designed for self-testing can identify people with previously unrecognized AF, this study may contribute to change the approach to screening for AF in the community. Consequently, the study may prevent stroke in the future. By preventing stroke, major personal and socio-economic consequences can be avoided.

ELIGIBILITY:
Inclusion Criteria:

* Age >65 years
* Diabetes, heart failure, hypertension, previous stroke/TIA or other cardiovascular disease (minimum 1 risk factor)
* Informed written consent for participation

Exclusion Criteria:

* Chronic AF
* Lack of ability to cooperate

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1500 (Actual)
Dates: Start 2020-12-23 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of AF | During procedure
  AF during procedure

CONTACTS AND LOCATIONS:
Overall Officials: Jarle Jortveit, PhD, Principal Investigator — Sorlandet Hospital Arendal
Locations (1):
- Sorlandet Hospital, Arendal, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sandberg EL, Halvorsen S, Berge T, Grimsmo J, Atar D, Leangen Grenne B, Jortveit J. Digital recruitment and compliance to treatment recommendations in the Norwegian Atrial Fibrillation self-screening pilot study. Eur Heart J Digit Health. 2024 Apr 9;5(3):371-378. doi: 10.1093/ehjdh/ztae026. eCollection 2024 May. PMID 38774377
- [Derived] Sandberg EL, Halvorsen S, Berge T, Grimsmo J, Atar D, Grenne BL, Jortveit J. Screening for Atrial Fibrillation by Digital Health Technology in Older People in Homecare Settings: A Feasibility Trial. Int J Telemed Appl. 2024 Mar 25;2024:4080415. doi: 10.1155/2024/4080415. eCollection 2024. PMID 38567031
- [Derived] Jortveit J, Boskovic M, Sandberg EL, Vegsundvag J, Halvorsen S. High Diagnostic Accuracy of Long-Term Electrocardiogram Interpretation by General Practitioners. Int J Telemed Appl. 2024 Feb 22;2024:6624344. doi: 10.1155/2024/6624344. eCollection 2024. PMID 38425473
- [Derived] Sandberg EL, Halvorsen S, Berge T, Grimsmo J, Atar D, Fensli R, Grenne BL, Jortveit J. Fully digital self-screening for atrial fibrillation with patch electrocardiogram. Europace. 2023 May 19;25(5):euad075. doi: 10.1093/europace/euad075. PMID 36945146
- [Derived] Jortveit J, Fensli R. Remote ECG Monitoring by ECG247 Smart Heart Sensor. Int J Telemed Appl. 2022 Feb 11;2022:6812889. doi: 10.1155/2022/6812889. eCollection 2022. PMID 35186075
- [Derived] Sandberg EL, Grenne BL, Berge T, Grimsmo J, Atar D, Halvorsen S, Fensli R, Jortveit J. Diagnostic Accuracy and Usability of the ECG247 Smart Heart Sensor Compared to Conventional Holter Technology. J Healthc Eng. 2021 Nov 2;2021:5230947. doi: 10.1155/2021/5230947. eCollection 2021. PMID 34765102
- See also: Related Info — http://www.afstudien.no